CLINICAL TRIAL: NCT04834505
Title: Construction and Validation of a Diagnosis Model Based on Endoscopic Ultrasound Characteristics for Differentiating Between Focal Autoimmune Pancreatitis and Pancreatic Cancer
Brief Title: To Differentiate Focal Autoimmune Pancreatitis From Pancreatic Cancer by Endoscopic Ultrasound
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Tao Guo, Associated professor in Department of Gastroenterolgy, Peking Union Medical College Hospital
Other Study IDs: EUS-AIP-PC-1
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Pancreatitis; Pancreatic Cancer
MeSH Terms: conditions — Autoimmune Pancreatitis; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation sample: The patients conclusively diagnosed as FAIP or PC are retrospectively collected.
  Interventions: Other: EUS for derivation sample
- Validation sample: The patients with difficulty in distinguishing between FAIP and PC are prospectively enrolled.
  Interventions: Other: Diagnostic imaging modalities for validation sample

INTERVENTIONS:
Other: Diagnostic imaging modalities for validation sample — Endoscopic ultrasound and other imaging modalities such as CT, MRI, or PET-CT are performed.
  Groups: Validation sample
Other: EUS for derivation sample — Endoscopic ultrasound was performed.
  Groups: Derivation sample

SUMMARY:
Autoimmune pancreatitis (AIP) is a special type of chronic pancreatitis mediated by autoimmunity. The classic manifestation of AIP is diffuse pancreatic enlargement, some of which are characterized by focal enlargement. Clinically, it is divided into diffuse AIP (DAIP) and focal AIP (FAIP) according to morphology. FAIP can be clinically manifested as obstructive jaundice, peripancreatic lymphadenopathy and vascular involvement, which may mimic pancreatic cancer (PC). CT/MRI is the important imaging tool for diagnosing pancreatic diseases. However, due to the overlap of the imaging features of FAIP and PC, it is challenging to differentiate the two by CT/MRI. Endoscopic ultrasound (EUS) can clearly display the pancreatic parenchyma and pancreatic duct system and has become a routine modality for the evaluation of pancreatic diseases. The aim of this study is to construct a diagnosis model for distinguishing between FAIP and PC by comparing the EUS characteristics of the two, and further validate its diagnostic efficacy.

DETAILED DESCRIPTION:
A derivation sample is established by retrospectively collecting the EUS images of about 100 FAIP patients and about 200 PC patients who were diagnosed for the first time in Peking Union Medical College Hospital in the past 6 years and underwent EUS at the same time. The parenchymal and ductal changes of pancreas were defined according to the Rosemont criteria. The parenchymal characteristics included hyperechoic foci/strands and lobularity, and the ductal changes included main pancreatic duct (MPD) dilation. Other EUS characteristics not included in the conventional criteria were described based on the literatures, including pancreatic diffuse hypoechogenicity, focal hypoechogenicity, pancreatic diffuse enlargement, focal enlargement, peripancreatic hypoechoic margin, common bile duct (CBD) dilation, bile duct wall thickening, lymphadenopathy and vessel involvement. The EUS characteristics of the two groups of patients are included in the multivariate stepwise logistic regression and receiver operating characteristics (ROC) analyses to construct a differential diagnosis model in derivation sample. Further, the differential diagnosis model will be prospectively validated by calculating the sensitivity and specificity in about 90 patients who are going to undergo EUS due to the difficulty in distinguishing between FAIP and PC. Diagnosis of AIP meets the revised Mayo clinic criteria (revised HISORt criteria) including features of histology, imaging, serology, other organs involvement and response to steroid therapy. Diagnosis of pancreatic duct adenocarcinoma is confirmed by surgical pathology or by cytology/histology after EUS-guided fine needle aspiration or biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with difficulty in distinguishing between FAIP and PC

Exclusion Criteria:

* Referred patients with a history of having being conclusively diagnosed as AIP or PC; Patients with DAIP; Patients with alcoholic pancreatitis, hypertriglyceridemia pancreatitis or pancreatitis due to gallstones; Patients with pancreatic cystic tumors, pancreatic neuroendocrine tumors or solid pseudopapillary tumors of pancreas; Patients who cannot undergo EUS due to unsuitable conditions.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In derivation sample, the patients conclusively diagnosed as FAIP or PC are retrospectively collected.
  In validation sample, the patients with difficulty in distinguishing between FAIP and PC are prospectively enrolled. In the end, the patient with a diagnosis that is neither FAIP nor PC and the patient without conclusive diagnosis are withdrawn from the study.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To construct a diagnosis model for distinguishing FAIP from PC and further validate its efficacy | 1 week after the diagnosis is conclusive
  Score is assigned to each predictor based on the odd ratio (OR) value, individual risk is estimated based on the sum of weighted score for each predictor and optimal cut-off point is obtained based on receiver operating characteristic (ROC) analysis.
  Sensitivity and specificity were used to assess the diagnostic efficacy.

SECONDARY OUTCOMES:
Compare the efficacy of EUS based on the model with that of CT/MRI/PET-CT in differentiating between FAIP and PC | 1 week after the diagnosis is conclusive
  Sensitivity and specificity were used to assess the diagnostic efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Tao Guo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The protocol of the study is private.

REFERENCES:
- [Background] Hart PA, Zen Y, Chari ST. Recent Advances in Autoimmune Pancreatitis. Gastroenterology. 2015 Jul;149(1):39-51. doi: 10.1053/j.gastro.2015.03.010. Epub 2015 Mar 12. PMID 25770706
- [Background] Kamisawa T, Okamoto A. Autoimmune pancreatitis: proposal of IgG4-related sclerosing disease. J Gastroenterol. 2006 Jul;41(7):613-25. doi: 10.1007/s00535-006-1862-6. PMID 16932997
- [Background] Miyabe K, Zen Y, Cornell LD, Rajagopalan G, Chowdhary VR, Roberts LR, Chari ST. Gastrointestinal and Extra-Intestinal Manifestations of IgG4-Related Disease. Gastroenterology. 2018 Oct;155(4):990-1003.e1. doi: 10.1053/j.gastro.2018.06.082. Epub 2018 Sep 12. PMID 30012334
- [Background] Muhi A, Ichikawa T, Motosugi U, Sou H, Sano K, Tsukamoto T, Fatima Z, Araki T. Mass-forming autoimmune pancreatitis and pancreatic carcinoma: differential diagnosis on the basis of computed tomography and magnetic resonance cholangiopancreatography, and diffusion-weighted imaging findings. J Magn Reson Imaging. 2012 Apr;35(4):827-36. doi: 10.1002/jmri.22881. Epub 2011 Nov 8. PMID 22069025
- [Background] Gardner TB, Levy MJ. EUS diagnosis of chronic pancreatitis. Gastrointest Endosc. 2010 Jun;71(7):1280-9. doi: 10.1016/j.gie.2010.02.038. No abstract available. PMID 20598255
- [Background] Hoki N, Mizuno N, Sawaki A, Tajika M, Takayama R, Shimizu Y, Bhatia V, Yamao K. Diagnosis of autoimmune pancreatitis using endoscopic ultrasonography. J Gastroenterol. 2009;44(2):154-9. doi: 10.1007/s00535-008-2294-2. Epub 2009 Feb 13. PMID 19214678
- [Background] Chari ST, Takahashi N, Levy MJ, Smyrk TC, Clain JE, Pearson RK, Petersen BT, Topazian MA, Vege SS. A diagnostic strategy to distinguish autoimmune pancreatitis from pancreatic cancer. Clin Gastroenterol Hepatol. 2009 Oct;7(10):1097-103. doi: 10.1016/j.cgh.2009.04.020. Epub 2009 May 4. PMID 19410017